CLINICAL TRIAL: NCT06377683
Title: An Open-Label, Non-Randomized, Single-Center, Investigator-Initiated Trial to Determine the Safety, Dosimetry, and Preliminary Effectiveness of 177Lu-Dansyl-PSMA in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Clinical Evaluation of 177Lu-DansyI-PSMA (LNC1011) in Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMYY-2023KY122
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Castration-resistant Prostate Cancer, mCRPC
Keywords: mCRPC; radioligand therapy; PSMA; 177Lu-DansyI-PSMA

STUDY DESIGN:
Intervention Model Description: classic 3+3 dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 177Lu-Dansyl-PSMA (Experimental): 177Lu-Dansyl-PSMA A maximum of 2 cycles of 50 mCi (1.85 GBq) 177Lu-Dansyl-PSMA, each. Route of administration: Slow intravenous infusion/injection (i.v.) Duration of treatment: 2 cycles, every 6 weeks. Subsequent cohorts received an incremental 50% dose increase until dose-limiting toxicity (DLT) was observed.
  Interventions: Drug: 177Lu-Dansyl-PSMA radioligand therapy

INTERVENTIONS:
Drug: 177Lu-Dansyl-PSMA radioligand therapy — Radioligand therapy using 177Lu-Dansyl-PSMA 50mCi (1.85GBq) will performed 6-weekly. A maximum of 2 cycles will be administered, and subsequent cohorts receive an incremental 50% dose increase until dose-limiting toxicity (DLT) was observed.

SUMMARY:
Ten to 20% of patients with prostate cancer (PC) experience progression in their disease, even after undergoing pharmaceutical or surgical castration, leading to metastatic CRPC (mCRPC). Prostate-specific membrane antigen (PSMA) is a membrane-bound glycoprotein mostly specific to the prostate. While PSMA is expressed at low levels in normal prostate, this expression increased by 100-1000-fold in PC, which makes it a favorable target for therapy. This study was designed to evaluate the safety, tolerability, and maximum tolerated dose of a long-lasting radiolabeled ligand 177Lu-Dansyl-PSMA in mCRPC patients.

DETAILED DESCRIPTION:
This proposal is a phase I, open-label study of escalating doses of 177Lu-Dansyl-PSMA Injection in patients with PSMA-positive mCRPC. The initial dose of 177Lu-Dansyl-PSMA is 1.85GBq (50 mCi), and subsequent cohorts receive an incremental 50% dose increase until dose-limiting toxicity (DLT) is observed. Treatment is planned for up to 2 cycles, and the time interval between cycles is 6 weeks. The primary endpoint assessed the safety and maximum tolerated dose of 177Lu-Dansyl-PSMA used for radioligand therapy in patients with PSMA-positive mCRPC. Secondary endpoints included dosimetry and determination of the preliminary treatment efficacy of 177Lu-Dansyl-PSMA.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign a written informed consent document.
2. Age 21 and older
3. Confirmed unresectable PC that is refractory to or has progressed following prior treatments.
4. Confirmed unresectable PC with measurable disease per RECIST (version 1.1) (i.e. at least 1 lesion > 1 cm or lymph node > 1.5 cm in short axis)
5. Patients must have a castrate level of serum/plasma testosterone (< 50 ng/dL or < 1.7 nmol/L).
6. Eastern Cooperative Oncology Group Performance Status ≤ 3
7. Participant must have completed prior therapy at least 2 weeks (washout period) before 68Ga-PSMA PET/CT scan. Any clinically significant toxicity (with the exceptions of hair loss and sensory neuropathy) related to prior therapy resolved below Grade 2 or baseline. Completion of entry into 68Ga-PSMA study and completion of the scan
8. Patients must be 68Ga-PSMA PET/CT scan positive.
9. Hematologic parameters defined as:

Absolute neutrophil count (ANC) ≥ 1000 cells/mm3 Platelet count ≥ 50,000/mm3 Hemoglobin ≥ 8 g/dL

Blood chemistry levels defined as:

AST, ALT, alkaline phosphatase ≤ 5 times upper limit of normal (ULN) Total bilirubin ≤ 3 times ULN Creatinine ≤ 3 times ULN Able to remain motionless for up to 30-60 minutes per scan

Exclusion Criteria:

1. Participant on any chemical anticoagulant including antiplatelet agents (excluding ASA)
2. Participants with Class 3 or 4 NYHA Congestive Heart Failure
3. Clinically significant bleeding within two weeks before trial entry (e.g. gastrointestinal bleeding, intracranial bleeding)
4. Major surgery, defined as any surgical procedure that involves general anesthesia and a significant incision (i.e. larger than what is required for placement of a central venous access, percutaneous feeding tube, or biopsy) within 28 days before study day 1 or anticipated surgery within the subsequent 6 weeks
5. Has an additional active malignancy requiring therapy within the past 2 years
6. Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
7. Psychiatric illness/social situations that would interfere with compliance with study requirements
8. Cannot undergo PET/CT scanning because of weight limits (350 lbs)
9. INR>1.2; PTT>5 seconds above UNL

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events (safety and tolerability) | At the end of Cycle 2 (each cycle is 42 days)
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. Dose-limiting toxicity was defined as any 177Lu-Dansyl-PSMA-related AE ≥ grade 3 (G3).
To determine the maximum tolerated dose (MTD) | At the end of Cycle 2 (each cycle is 42 days)
  The MTD is the dose level below that which 2 out of 6 subjects in a cohort have DLT

SECONDARY OUTCOMES:
Dosimetry | At the end of Cycle 1 (each cycle is 42 days)
  Dosimetry, measured as absorbed dose in tumor and normal organs (Gy/GBq), was estimated in the first treatment cycle for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Haojun Chen, MD, PhD, Study Chair — The First Affiliated Hospital of Xiamen University
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China